CLINICAL TRIAL: NCT01456689
Title: A Multi-Center, Open-Label, Dose Escalation, Phase 1 Study of Oral LGH447 in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of Oral LGH447 in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLGH447X2101; 2011-003820-10 (EudraCT Number)
Record Dates: First submitted 2011-10-11; First posted 2011-10-21 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; MM
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — LGH-447; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LGH447 (Experimental): Eligible patients will be treated with oral LGH447 until disease progression or occurrence of unacceptable toxicity.
  Interventions: Drug: LGH447
- LGH447 and midazolam (Experimental): Eligible patients will receive midazolam on two separate days, the first dose will be administered prior to the start of LGH447 and the second will be co-administered with LGH447. After that, the patients will continue to be treated with oral LGH447 until disease progression or occurrence of unacceptable toxicity.
  Interventions: Drug: LGH447; Drug: midazolam

INTERVENTIONS:
Drug: LGH447
Drug: midazolam
  Arms: LGH447 and midazolam

SUMMARY:
The primary purpose of this dose escalation study is to estimate the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) of LGH447 as a single agent when administered orally once daily to adult patients with Multiple Myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma that is relapsed and/or refractory for which no curative option exists.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* During the dose expansion part of the study patients must have measurable disease defined by at least 1 of the following 2 measurements:

  * Serum M-protein ≥ 0.5 g/dL
  * Urine M-protein ≥ 200 mg/24 hours
  * Serum free light chain (FLC) > 100 mg/L of involved FLC

Exclusion Criteria:

* Patients who are currently receiving treatment with medications that meet one of the following criteria and that cannot be discontinued at least one week prior to the start of treatment with LGH447:

  * Strong inhibitors or inducers of CYP3A4
  * CYP3A4 substrates with narrow therapeutic index

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-04-25 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Estimate the MTD and/or RDE | 12 months
  Incidence rate of dose limiting toxicity

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events. | 18 months
  Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Pharmacokinetic (PK) effects of LGH447 | 18 months
  Summary of PK parameters such as AUC, Cmax,
Pharmacodynamic (PD) effects of LGH447 | 18 months
  Changes between pre and post treatment levels in bone marrow aspirates and whole blood.
Anti-Myeloma activity associated with LGH447 | 18 months
  Overall Response Rate (ORR), Duration of Response (DOR), and Progression Free Survival (PFS) based on International Myeloma Working Group Response Criteria.
Effect of multiple-doses of LGH447 on the PK of midazolam | 6 months
  PK parameters of midazolam and 1-hydroxymidazolam, such as AUC and Cmax, as well as metabolic ratio of midazolam.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (4):
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Houston, Texas
- Germany (2):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLGH447X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17667